CLINICAL TRIAL: NCT00867828
Title: Multi-Center, Double-Blind, Placebo-Controlled, Monotherapy Study of Neptune Krill Oil (NKO™) in Early Stage Alzheimer's Disease
Brief Title: Neptune Krill Oil (NKO™) in Early Stage Alzheimer's Disease (MNEMOSYNE)
Acronym: MNEMOSYNE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NeuroBioPharm Inc. (Industry)
Collaborators: Neptune Technologies and Bioressources Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBP-4209AD; NCT00861289 (obsolete NCT alias)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Early Onset Alzheimer Disease
Keywords: Decline of global cognitive function; Neuropsychological Test Battery (NTB); Early stage Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Neptune Krill Oil(TM)softgels (1g QD). Each softgel of Neptune Krill Oil will provide approximately 150 mg EPA and 100 mg DHA.
  Interventions: Dietary Supplement: Neptune Krill Oil
- 2 (Active Comparator): Fish oil softgels (1g QD). Each softgel of Fish Oil will provide approximately 150 mg EPA and 100 mg DHA.
  Interventions: Dietary Supplement: Fish Oil
- 3 (Placebo Comparator): Placebo (soy oil) softgels (1g QD. The soy oil placebo will provide neither EPA nor DHA.
  Interventions: Dietary Supplement: Placebo (soy oil)

INTERVENTIONS:
Dietary Supplement: Neptune Krill Oil — Softgels 1g QD. Each softgel of Neptune Krill Oil will provide approximately 150 mg EPA and 100 mg DHA.
  Arms: 1
Dietary Supplement: Fish Oil — Softgels 1g QD. Each softgel of Fish Oil will provide approximately 150 mg EPA and 100 mg DHA.
  Arms: 2
Dietary Supplement: Placebo (soy oil) — Softgels 1g QD. The soy oil placebo will provide neither EPA nor DHA.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy of NKO™ softgels in reducing decline of global cognitive function as measured by the Neuropsychological Test Battery (NTB), in patients diagnosed with early stage Alzheimer's disease when compared to fish oil and a placebo after 24 weeks of treatment.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is an irreversible, progressive neurodegenerative disorder, characterized by gradual cognitive deterioration, changes in behavior and personality. These symptoms are related to neurochemical changes, neural death, and the breakdown of the inter-neural connections. Loss of short-term memory is often the first sign, followed by cognitive deficits involving multiple functions. Early stages of AD and mild cognitive impairment are characterized as milder forms of memory loss or cognitive impairment that could precede the onset of dementia and AD. Prevention of further cognitive decline inpatients with these possible precursor conditions is of paramount importance given that reversibility of AD is not possible.

It is estimated there are currently about 5.1 million people with Alzheimer's disease (AD) in the United States (Alzheimer's Association, 2007) and this number is expected to reach 13.2 millions by 2050 (Hebert et al., 2003). Alzheimer's is ranked as the 7th leading cause of death in the US for people of all ages and the 5th for people aged 65 or older (National Center for Health Statistics, 2004). In Canada it is 280,000 people over 65 that are estimated to have AD, and over 750,000 are expected to have the disease by 2031 (Alzheimer Society of Canada, 2006). It is estimated to 10% of all North Americans over the age of 70 years have early stage AD or mild cognitive impairment.

Older age, low educational level and APOE ε4 allele are risk factors for AD (Lindsay et al., 2002). Moreover, patients having the APOE ε4 allele show an earlier and faster cognitive decline while having the ε2 allele is related to a slower decline. Homozygotous ε4 patients show an even earlier and faster decline than heterozygotes (Martins et al., 2005).

While symptomatic treatments have been the focus of therapeutic investigations for AD, recent research efforts target the toxic effect of amyloid beta (Aβ) peptides in order to modify the underlying pathophysiology of the disease.

The presently approved treatments give only small clinical improvement and do not prevent the progression of the disease, from mild cognitive impairment to dementia and death (Birks et al., 2000; AD2000 Collaborative Group, 2004; Birks, 2006; Birks & Harvey, 2006; Loy & Schneider, 2006).

Alzheimer's disease is characterized by two main pathological features of the brain: intracellular neurofibrillary tangles formed by abnormal protein τ (tau); and extracellular neuritic plaques formed by β-amyloid peptides (Aβ) (Kuo et al., 1996). The overproduction of Aβ42 is genetically induced but environmental risk factors are required to get fully symptomatic AD (Grant et al., 2002).

Among these risk factors, low docosahexaenoic acid (DHA) is one of the most important dietary risk factor for AD (Morris et al., 2005). The reasons for the impact of DHA on learning and memory and the association with AD are unclear but could result from its loss in synapses (Montine et al., 2004), which are normally rich in DHA (Salem et al., 2001), where it is particularly important for postsynaptic transmission and neuroprotection (Bazan, 2003). Studies in animal models have consistently showed that brain n-3 fatty acid content is highly dependent on dietary intake and aging (Favrere et al., 2000; Youdim et al., 2000; Calon & Cole, 2007).

Several animal studies, has shown that increased DHA intake has been found to increase hippocampal acetycholine levels and its derivatives, neuroprotectin DI, which deceased cell death (Aid et al, 2005; Lukiw et al., 2005). A study conducted on aged mice showed that DHA intake improved memory performance (Lim et al. 2001). In another Alzheimer's disease mouse model, reduction in dietary DHA showed loss of postsynaptic proteins associated with increased oxidation, which was localized in the dendrites. However, when a group of DHA-restricted mice where given DHA, they showed signs that the DHA intake protected them against dendritic pathology, implying that DHA could be useful in preventing cognitive impairment in Alzheimer's Disease (Calon et al., 2004).

Several epidemiological studies have shown a protective effect associated with increased fish intake (a direct source of omega 3 fatty acids) against dementia and cognitive impairment decline (Kalmijin et al. 1997, Barberger-Gateau et al. 2002; Morris et al 2003). Recently, one large randomized double-blind placebo-controlled study found 1.6 g DHA and 0.7 EPA may be beneficial in reducing risk for AD (Freund-Levi et al, 2006). In addition, there is mounting evidence that dietary supplementation with Omega 3 Fatty acids may be beneficial in different psychiatric conditions such as mood behaviour, depression and dementia (Bourre et al., 2005; Peet and Stokes, 2005; Stoll et al., 1999).

Krill is a very small crustacean which thrives in deep cold ocean waters where it forms an important part of the life chain, providing nutrition for an array of marine mammals, birds and fish. Neptune Krill oil (NKO) is a rich source of omega-3 and omega-9 fatty acids and phospholipids, which carry and thus functionalize the omega-3 fatty acids (EPA/DHA) attached. Phospholipids are important in protecting membranes from toxic injury and free radical attack (Everson, I et al. 2000). NKO contains two main potent antioxidants; a carotenoid (astaxanthin) and a flavonoid (novel due to its animal source). Astaxanthin has been shown to have a stronger antioxidant activity than alpha-tocopherol, beta-carotene, lycopene and lutein. Flavonoids, traditionally extracted from fruits, plants, vegetables or algae have been studied for more than 60 years and their antioxidant activity is undoubted.

The hypothesis that NKO will be effective in AD is based on the high content of phospholipids with DHA and of antioxidants that cross the blood - brain barrier as well as essential brain nutrients. In addition, NKO has been proven to increase HDL-C that is related to decreased plague formation which is related to decreased blood supply to the brain, one of the factors causing AD progression. The aim of the current study is to challenge this hypothesis in a randomized double blind study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years or older.
* Patients with a clinical diagnosis of early stage Alzheimer's disease (NINCDS-ADRDA criteria) and with a Standardized Mini-Mental State Examination (MMSE) score of 20 - 26 inclusively and have demonstrated decline in their cognitive functions during the last six months as determined by the treating physicians.
* Patient has a score < 9 on the Hamilton Rating Scale for Depression (Ham-D) (Vida et al., 1994; Naarding et al., 2002).
* If on anti-depressant treatment and/or treatment for any other psychiatric condition the dose must have been stable for six months prior to randomization and should continue to be on the same stable dose for the entire treatment duration.
* Patient is not taking fish oil or Omega 3/6 supplement 2 weeks before screening visit.
* Patient is living at home or in a home for elderly persons.
* Patient has a responsible caregiver who is able to provide information about the patient's functional status.
* If on a cholinesterase inhibitor treatment the dose must have been stable for at least six months prior to randomization and should continue to be on the same stable dose for the entire treatment duration.
* If on any concomitant medication treatment the dose must have been stable for at least four months prior to randomization and should continue to be on the same stable dose for the entire treatment duration.
* Written informed consent is obtained from the patient or the legally accepted representative.

Exclusion criteria:

* Women who are pregnant or with childbearing potential and not willing to take adequate birth control measures.
* Severe or unstable diseases of any type, other than cognitive impairment, that may interfere with outcome evaluations. These include medical conditions expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical or mental status of the patient to a significant degree or put the patient at special risk.
* Intake of fish oil or Omega 3/6 supplement other than the study drug
* Patients are taking more than 400 mg vitamin E.
* The patient is not able to reliably take the study medication for the duration of the study (Patient compliance is < 60% after the 2-week run-in period).
* Patients with severe medical condition(s) that in the view of the treating physician prohibits participation in the study.
* Patients using any other investigational agent, or participating in another study within the last 30 days prior to the baseline visit.
* Patient with known allergy to fish, seafood or soy/soy-derived products.
* Patient diagnosed with coagulopathy or on anticoagulant therapy
* Patient subject to symptomatic hypoglycemia.
* Patient requires to be initiated on an anti-depressant medication and/or treatment for any other psychiatric condition prior to randomization.
* Patient requires to be initiated on a cholinesterase inhibitor treatment prior to randomization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change in Neurological Test Battery between baseline and 24 weeks of treatment. | Between baseline and 24 weeks of treatment

SECONDARY OUTCOMES:
Secondary outcome measures will include the change in DAD at 24 weeks of treatment, the change in NTB, GDS, DAD, and MMSE at 12 weeks.Safety and tolerability will be assessed by the incidence of treatment emergent adverse events. | 24 week period

CONTACTS AND LOCATIONS:
Locations (14):
- Canada (14):
  - Surrey, British Columbia
  - Deer Lake, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Cornwall, Ontario
  - Hamilton, Ontario
  - Hawkesbury, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Thornhill, Ontario
  - Thunder Bay, Ontario
  - Dollard-des-Ormeaux, Quebec
  - Grand-Mère, Quebec
  - Montreal, Quebec